CLINICAL TRIAL: NCT00774137
Title: Phase IV Multi Center Validation Study of Novel Biomarkers of Acute Kidney Injury After Cardiac Surgery
Brief Title: Examining New Diagnostic Tests for Acute Kidney Injury After Heart Surgery
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0603001221; R01HL085757 (NIH)
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Kidney Failure, Acute; Renal Insufficiency
Keywords: Acute Kidney Injury; IL-18; NGAL; Cystatin C; Biomarkers; Dialysis
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, plasma, buffy coat (optional)
Oversight: Data Monitoring Committee: No

SUMMARY:
People who undergo coronary artery bypass grafting (CABG) or heart valve surgery may experience acute kidney injury (AKI) after their surgery. Current medical tests cannot identify AKI until approximately 48 hours after it occurs. This study will examine three new biomarkers in blood and urine that may provide a more effective and faster way of predicting AKI in people who undergo CABG or heart valve surgery.

DETAILED DESCRIPTION:
AKI, which is indicated by a sudden change in serum creatinine levels, is a serious complication that can occur after a patient undergoes CABG or heart valve surgery. People who experience AKI after heart surgery may be at increased risk for post-operative complications, including long-term kidney failure or heart damage. AKI is currently identified by testing serum creatinine levels in the blood, which is the traditional marker of kidney function. However, serum creatinine levels can be affected by other non-kidney-related factors and may not positively identify AKI until 48 hours after it begins. This study will examine three new biomarkers found in urine and blood-urine interleukin 18 (IL-18), neutrophil gelatinase-associated lipocalin (NGAL), and cystatin C-that may be able to predict AKI more effectively and faster than serum creatinine levels. In addition, study researchers will also determine if changes in these biomarkers can predict the severity of AKI more successfully than serum creatinine tests.

This study will enroll people undergoing CABG or heart valve surgery at Yale-New Haven Hospital. Before the surgery and once a day for 5 days after the surgery, blood and urine collection will occur. Study researchers will also review participants' medical records. Twelve months after hospital discharge, participants will return to the clinic for a follow-up visit for repeat blood and urine collection and to complete questionnaires. A portion of blood will be saved for future genetic testing; this is optional.

ELIGIBILITY:
Inclusion Criteria for Adults: (must have at least one of the following)

* Emergent surgery
* Pre-existing kidney impairment (baseline serum creatinine greater than 2 mg/dL)
* Ejection fraction less than 35%
* At least 70 years old
* Diabetes mellitus
* Combined CABG and valve surgery
* Repeat CABG or valve surgery

Exclusion Criteria for Adults:

* Pre-operative acute kidney injury
* Enrolled in a conflicting research study
* Prior kidney transplantation
* Baseline serum creatinine level greater than 4.5 mg/dL
* Nephrotoxic drugs administered pre-operatively
* Surgery for only left ventricular assist device

Inclusion Criteria for Children:

* Undergoing open heart surgery

Exclusion Criteria for Children:

* Pre-existing acute kidney failure (greater than 50% decline in creatinine clearance)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Adults undergoing CABG surgery or heart valve surgery.
  2. Children undergoing cardic surgery (requiring CABG) to correct congenital heart defects.
Sampling Method: Non-Probability Sample
Enrollment: 1550 (Actual)
Dates: Start 2007-04; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Changes in serum creatinine levels (absolute and percentage) | Measured in the 1 week after surgery

SECONDARY OUTCOMES:
Doubling of serum creatinine, use of dialysis, or death | Measured during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Chirag R. Parikh, MD, PhD, Principal Investigator — Yale University
Locations (8):
- United States (6):
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Chicago School of Medicine, Chicago, Illinois
  - Duke Clinical Research Institute, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Montreal Children's Hospital at McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Result] Parikh CR, Coca SG, Thiessen-Philbrook H, Shlipak MG, Koyner JL, Wang Z, Edelstein CL, Devarajan P, Patel UD, Zappitelli M, Krawczeski CD, Passik CS, Swaminathan M, Garg AX; TRIBE-AKI Consortium. Postoperative biomarkers predict acute kidney injury and poor outcomes after adult cardiac surgery. J Am Soc Nephrol. 2011 Sep;22(9):1748-57. doi: 10.1681/ASN.2010121302. Epub 2011 Aug 11. PMID 21836143
- [Result] Li S, Krawczeski CD, Zappitelli M, Devarajan P, Thiessen-Philbrook H, Coca SG, Kim RW, Parikh CR; TRIBE-AKI Consortium. Incidence, risk factors, and outcomes of acute kidney injury after pediatric cardiac surgery: a prospective multicenter study. Crit Care Med. 2011 Jun;39(6):1493-9. doi: 10.1097/CCM.0b013e31821201d3. PMID 21336114
- [Result] Parikh CR, Devarajan P, Zappitelli M, Sint K, Thiessen-Philbrook H, Li S, Kim RW, Koyner JL, Coca SG, Edelstein CL, Shlipak MG, Garg AX, Krawczeski CD; TRIBE-AKI Consortium. Postoperative biomarkers predict acute kidney injury and poor outcomes after pediatric cardiac surgery. J Am Soc Nephrol. 2011 Sep;22(9):1737-47. doi: 10.1681/ASN.2010111163. Epub 2011 Aug 11. PMID 21836147
- [Result] Shlipak MG, Coca SG, Wang Z, Devarajan P, Koyner JL, Patel UD, Thiessen-Philbrook H, Garg AX, Parikh CR; TRIBE-AKI Consortium. Presurgical serum cystatin C and risk of acute kidney injury after cardiac surgery. Am J Kidney Dis. 2011 Sep;58(3):366-73. doi: 10.1053/j.ajkd.2011.03.015. Epub 2011 May 20. PMID 21601336
- [Result] Zappitelli M, Krawczeski CD, Devarajan P, Wang Z, Sint K, Thiessen-Philbrook H, Li S, Bennett MR, Ma Q, Shlipak MG, Garg AX, Parikh CR; TRIBE-AKI consortium. Early postoperative serum cystatin C predicts severe acute kidney injury following pediatric cardiac surgery. Kidney Int. 2011 Sep;80(6):655-62. doi: 10.1038/ki.2011.123. Epub 2011 Apr 27. PMID 21525851
- [Derived] Kavsak PA, Belley-Cote EP, Whitlock RP, Lamy A. Cardiac troponin testing in cardiac surgery. Expert Rev Cardiovasc Ther. 2023 Jul-Dec;21(11):729-731. doi: 10.1080/14779072.2023.2283123. Epub 2023 Dec 10. No abstract available. PMID 37947177
- [Derived] Menez S, Ju W, Menon R, Moledina DG, Thiessen Philbrook H, McArthur E, Jia Y, Obeid W, Mansour SG, Koyner JL, Shlipak MG, Coca SG, Garg AX, Bomback AS, Kellum JA, Kretzler M, Parikh CR; Translational Research Investigating Biomarker Endpoints in AKI (TRIBE-AKI) Consortium and the Kidney Precision Medicine Project. Urinary EGF and MCP-1 and risk of CKD after cardiac surgery. JCI Insight. 2021 Jun 8;6(11):e147464. doi: 10.1172/jci.insight.147464. PMID 33974569
- [Derived] Koyner JL, Garg AX, Thiessen-Philbrook H, Coca SG, Cantley LG, Peixoto A, Passik CS, Hong K, Parikh CR; TRIBE-AKI Consortium. Adjudication of etiology of acute kidney injury: experience from the TRIBE-AKI multi-center study. BMC Nephrol. 2014 Jul 4;15:105. doi: 10.1186/1471-2369-15-105. PMID 24996668
- [Derived] Hornik CP, Krawczeski CD, Zappitelli M, Hong K, Thiessen-Philbrook H, Devarajan P, Parikh CR, Patel UD; TRIBE-AKI Consortium. Serum brain natriuretic peptide and risk of acute kidney injury after cardiac operations in children. Ann Thorac Surg. 2014 Jun;97(6):2142-7. doi: 10.1016/j.athoracsur.2014.02.035. Epub 2014 Apr 13. PMID 24725832
- [Derived] Koyner JL, Garg AX, Coca SG, Sint K, Thiessen-Philbrook H, Patel UD, Shlipak MG, Parikh CR; TRIBE-AKI Consortium. Biomarkers predict progression of acute kidney injury after cardiac surgery. J Am Soc Nephrol. 2012 May;23(5):905-14. doi: 10.1681/ASN.2011090907. Epub 2012 Mar 1. PMID 22383693
- [Derived] Patel UD, Garg AX, Krumholz HM, Shlipak MG, Coca SG, Sint K, Thiessen-Philbrook H, Koyner JL, Swaminathan M, Passik CS, Parikh CR; Translational Research Investigating Biomarker Endpoints in Acute Kidney Injury (TRIBE-AKI) Consortium. Preoperative serum brain natriuretic peptide and risk of acute kidney injury after cardiac surgery. Circulation. 2012 Mar 20;125(11):1347-55. doi: 10.1161/CIRCULATIONAHA.111.029686. Epub 2012 Feb 9. PMID 22322531
- [Derived] Coca SG, Jammalamadaka D, Sint K, Thiessen Philbrook H, Shlipak MG, Zappitelli M, Devarajan P, Hashim S, Garg AX, Parikh CR; Translational Research Investigating Biomarker Endpoints in Acute Kidney Injury Consortium. Preoperative proteinuria predicts acute kidney injury in patients undergoing cardiac surgery. J Thorac Cardiovasc Surg. 2012 Feb;143(2):495-502. doi: 10.1016/j.jtcvs.2011.09.023. Epub 2011 Nov 3. PMID 22050987